CLINICAL TRIAL: NCT05726565
Title: Impact of Cardiac Rehabilitation on Acute Heart Failure Patients With Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200636B0
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure, Systolic; Morality; Cognitive Impairment
Keywords: acute heart failure; cognitive screening; cardiac rehabilitation; cardiopulmonary exercise test; adverse outcomes
MeSH Terms: conditions — Heart Failure, Systolic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LNNB-S >=10: As one of the core components of multidisciplinary CR, psychiatrist and psychologist consultation was delivered to all patients. Cognitive function was assessed with the Luria-Nebraska Neuropsychological Battery-Screening test (LNNB-S) Chinese version by an experienced psychologist. The evaluation would be completed during admission. The initial LNNB was condensed to fifteen items for the screen test by Golden. LNNB-S Chinese version focuses on 3 domains, including number calculation, cognitive function, and rhythm control. In our participants' cohort, investigators choose LNNB-S >=10 as a cutoff point. That is, participants may have cognitive impairment when their LNNB-S >=10.
  Interventions: Other: multidisciplinary cardiac rehabilitation
- LNNB-S <10: As one of the core components of multidisciplinary CR, psychiatrist and psychologist consultation was delivered to all patients. Cognitive function was assessed with the Luria-Nebraska Neuropsychological Battery-Screening test (LNNB-S) Chinese version by an experienced psychologist. The evaluation would be completed during admission. The initial LNNB was condensed to fifteen items for the screen test by Golden. LNNB-S Chinese version focuses on 3 domains, including number calculation, cognitive function, and rhythm control. In our participants' cohort, investigators choose LNNB-S >=10 as a cutoff point. That is, participants may have cognitive impairment when their LNNB-S >=10.
  Interventions: Other: multidisciplinary cardiac rehabilitation

INTERVENTIONS:
Other: multidisciplinary cardiac rehabilitation — A heart failure disease management program was delivered to all patients before discharge, including an HF specialist nurse education program, dietitian consultation, physiatrist consultation, and psychologist consultation and assessment. Participants were advised to receive phase II CR after the CPET within one month. Moderate continuous aerobic exercise training was prescribed individually according to the CPET result.4 The training intensity was within 10 beats of the anaerobic threshold or 40-60% of peak VO2. The training intensity was gradually increased fortnightly as tolerated (Borg's scale of 12-14). Phase II CR consisted of 12 weeks of 36 sessions in the entire course. Patients who received at least one exercise session were considered as receiving CR. Other patients were considered non-receiving CR.

SUMMARY:
In heart failure patients, neuropsychological disorders have been prospectively linked to frequent hospitalizations, recurrent cardiac events, and mortality. Cognitive dysfunction is also a frequent comorbidity in heart failure (HF) patients. The benefit of cardiac rehabilitation between patients with cognitive dysfunction and patients without cognitive dysfunction is unknown. Investigators hypothesize that patients with cognitive dysfunction benefit more from cardiac rehabilitation programs than patients without cognitive dysfunction.

DETAILED DESCRIPTION:
Investigators retrospectively reviewed HF patients discharged from acute HF hospitalizations between March 2015 and May 2021 at the heart failure center, Kaohsiung Chang Gung Memorial Hospital. Cognitive function was assessed with the Luria-Nebraska Neuropsychological Battery-Screening test (LNNB-S) Chinese version by an experienced psychologist. Participants may have cognitive impairment when their LNNB-S >=10. A heart failure disease management program was delivered to all patients before discharge, including an HF specialist nurse education program, dietitian consultation, physiatrist consultation, and psychologist consultation and assessment. Participants were advised to receive phase II cardiac rehabilitation (CR) after the cardiopulmonary exercise test (CPET) within one month. Moderate continuous aerobic exercise training was prescribed individually according to the CPET result. Participants who received at least one exercise session of phase II CR were considered as receiving CR. Other participants were considered non-receiving CR. Kaplan-Meier curves and log-rank test were constructed to compare the composite endpoint and all-causes mortality in four groups (Group a: Candidates without cognitive impairment and receiving CR. Group b: Candidates without cognitive impairment and not-receiving CR. Group c: Candidates with cognitive impairment and receiving CR. Group d: Candidates with cognitive impairment and not-receiving CR.)

ELIGIBILITY:
Inclusion Criteria:

* acute HF patients with reduced ejection fraction (left ventricular ejection fraction, LVEF <=40%) and discharged alive from the hospital.
* Completed cognitive and psychological functional assessment.
* Aged >= 20 years of age, male or female.
* Received heart failure disease management coordinated by an HF specialist nurse as described before.

Exclusion Criteria:

* Estimated survival time < 6 months.
* Long-term bedridden for more than 3 months.
* Terminal heart status. 4. Cannot cooperate with all functional studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators retrospectively reviewed 247 HF patients who were discharged from an acute HF hospitalization. LNNB-S was assessed in all patients. Multivariate Cox Regression by enter method was used to determine significant predictors for all-cause mortality and composite endpoints. Kaplan-Meier curves and log-rank test were constructed to compare the composite endpoint and all-causes mortality according to cognitive impairment and receiving CR.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
composite of all-cause mortality or HF hospitalization | March, 2015 ~ May, 2021
  Number of participants that had an occurrence of the mortality which is defined as all-cause mortality or occurrence of HF hospitalization

SECONDARY OUTCOMES:
all-cause mortality | March, 2015 ~ May, 2021
  Number of participants that had occurrence of the mortality which is defined as all-cause mortality
recurrent HF hospitalization | March, 2015 ~ May, 2021
  Number of participants that had an occurrence of HF hospitalization
Change From Baseline to Month 6 and Month 12 for the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ 12) Clinical Summary Score | March, 2015 ~ May, 2021
  Change from baseline to Month 6 and month 12 for the Kansas City Cardiomyopathy Questionnaire short form (KCCQ12) clinical summary score. KCCQ12 is a 12-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ12 clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital Heart Failure Center, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing plans will be discussed with other investigators